CLINICAL TRIAL: NCT00819520
Title: A Randomised, Double-Blind, Multicentre Study to Compare the Efficacy and Tolerability of Oral Ivermectin to Malathion 0.5% Lotion in the Treatment of Head Lice Infestation
Brief Title: Ivermectin in the Treatment of Head Lice
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 075-00
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2011-08-22 (Estimated); Status verified 2011-08

CONDITIONS: Lice Infestations
Keywords: pediculosis capitis; pediculus
MeSH Terms: conditions — Lice Infestations | interventions — Ivermectin; Malathion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ivermectin (Experimental): ivermectin Stromectol®)
  Interventions: Drug: ivermectin
- Malathion (Active Comparator): malathion(Prioderm®)
  Interventions: Drug: malathion

INTERVENTIONS:
Drug: ivermectin — Two single doses of oral ivermectin 400 mcg/kg (Days 1 and 8) plus 2 single applications of placebo lotion
  Other Names: Stromectol®
  Arms: Ivermectin
Drug: malathion — Two single applications of malathion 0.5% lotion (Days 1 and 8) plus 2 single doses of placebo tablets
  Other Names: Prioderm®
  Arms: Malathion

SUMMARY:
The purpose of this study is to compare 2 single doses of ivermectin as tablets with 2 single applications of malathion 0.5% lotion (Days 1 and 8) in clearing head lice, in patients who have recently used standard head lice treatments without success.

DETAILED DESCRIPTION:
Head lice infestation occurs frequently, primarily in children 3 to 11 years of age. In recent years an increasing prevalence of lice infestation in schools, day care centres, and summer day camps is believed to be partly due to increasing lice resistance to currently available standard treatments for pediculosis (infestation with lice). There is a need for new effective backup treatments for this common condition of head lice infestation. This is a double-blind, randomized, parallel-group, study in several clinical centres comparing ivermectin as tablets to malathion 0.5% lotion in the treatment of head lice. All enrolled patients participate in the primary phase of the study up to the Day 15 evaluation. Patients who are still infested with lice at Day 15 (treatment failures) will enter an extension phase and be treated in a double-blind, fashion with the opposite treatment (ie ivermectin or malathion). The study hypothesis is that ivermectin will be more effective than malathion in clearing head lice infestation , as measured by the proportion of patients who are lice-free at Study Day 15.

ELIGIBILITY:
Inclusion Criteria:

* Head lice infestation confirmed by detection combing by study staff
* previous (within 6 weeks) use of a topical insecticide product
* minimum 15kg weight
* providing informed consent

Exclusion Criteria:

* pregnant or nursing patients
* households with 7 or more infested patients
* households where there are other known infested household members not participating
* head lice treatment within 2 weeks of entry
* active scalp infection
* any difficulty with combing assessment
* patient from region endemic for certain parasitic worm diseases

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 812 (Actual)
Dates: Start 2004-02; Primary Completion 2004-09 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Absence or presence of live head lice | Study Day 15

SECONDARY OUTCOMES:
Absence or presence of live head lice at alternative Study Days. | Study Days 2, 8, 22, 29
Safety Assessments will consist of monitoring and recording all non-serious Adverse Events (AEs) and Serious Adverse Events (SAEs), their frequency, severity, seriousness, and relationship to the investigational product. | throughout duration of the study (+ 30 days for spontaneously reported SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Cottrell, Study Director — J&J Consumer and Personal Products Worldwide
Locations (4):
- Hopital Avicenne, Bobigny, Paris, France
- Shandon Clinic, Cork, Co. Cork, Ireland
- Chaim Sheba Medical Centre, Tel Litwinsky, Tel Hashomer, Israel
- Synexus Clinical Research Centre, Reading, Berks, United Kingdom

REFERENCES:
- [Derived] Chosidow O, Giraudeau B, Cottrell J, Izri A, Hofmann R, Mann SG, Burgess I. Oral ivermectin versus malathion lotion for difficult-to-treat head lice. N Engl J Med. 2010 Mar 11;362(10):896-905. doi: 10.1056/NEJMoa0905471. PMID 20220184